CLINICAL TRIAL: NCT05273164
Title: State Representation in Early Psychosis
Acronym: STEP
Status: Completed | Type: Observational
Sponsor: University of Minnesota (Other)
Collaborators: National Institute of Mental Health (NIMH) (NIH)
Responsible Party: Principal Investigator, Sophia Vinogradov, Professor and Department Head, University of Minnesota
Other Study IDs: STUDY00009964; 5P50MH119569 (NIH)
Record Dates: First submitted 2022-01-24; First posted 2022-03-10 (Actual); Last update posted 2025-09-22 (Actual); Status verified 2025-09

CONDITIONS: Psychosis; Schizophrenia; Schizophrenia Spectrum and Other Psychotic Disorders; Schizoaffective Disorder
MeSH Terms: conditions — Psychotic Disorders; Schizophrenia; Schizophrenia Spectrum and Other Psychotic Disorders

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | Unapproved Device: Yes | US Export: No

GROUPS / COHORTS (2):
- Early Psychosis participants: Individuals who have been diagnosed with a psychosis spectrum illness, such as schizophrenia, and are in the early stages of the disease (i.e., aged 15-35, or if 36-45, has had the onset of psychotic symptoms within the last 5 years)
- Healthy Controls: Demographically matched participants who do not have a personal or immediate family history of psychosis spectrum illnesses.

SUMMARY:
The purpose of this study is to examine state representation in individuals aged 15-45 who have been diagnosed with a psychotic illness, as well as young adults who do not have a psychiatric diagnosis. State Representation is our ability to process information about our surroundings. Participants will complete computerized tasks that measure state representation while having their brain activity measured.

DETAILED DESCRIPTION:
Participants will be asked to complete two sets of appointments six months apart. During both sets of appointments, participants will be asked to complete interviews examining behaviors and symptoms of mental health conditions, self-report questionnaires, and a neurocognitive assessment. In addition, participants will complete an imaging appointment, in which they will receive simultaneous electroencephalography (EEG) and functional Magnetic Resonance Imaging (fMRI) while performing two computerized tasks.

The purpose of this study is to determine how differences in information processing that support state representation in neural circuits relate to clinical heterogeneity in early psychosis. To this end, the investigators will: (a) Recruit people with early psychosis and demographically similar adults without a psychiatric illness aged 15-45 years; (b) Determine test-retest reliability of variants of the Dot Pattern Expectancy (DPX) and Bandit tasks as assessments of state representation processes; (c) Characterize behavioral performance and neurophysiology at baseline using the DPX and Bandit task variants during simultaneous EEG-fMRI along with other MRI modalities; (d) Follow patients for 6 months while they receive usual care, to delineate their clinical trajectories; (e) Repeat the behavioral and EEG-fMRI assessments after six months. The data the investigators acquire will allow us to examine the baseline relationships between clinical and experimental measures, and also to investigate how changes in clinical and experimental measures are related over a 6-month time period during a critical phase of illness.

Participants in this protocol will be invited to participate in a follow on study, NCT05664594.

ELIGIBILITY:
Inclusion Criteria:

* English proficiency, as determined by staff observation and participant self-report
* Estimated IQ at or above 70, as estimated by the cognitive assessments

Additional Inclusion Criteria for Early Psychosis Participants:

* Clinical diagnosis of schizophrenia, schizoaffective disorder, schizophreniform disorder, psychosis NOS, bipolar disorder with psychosis, or major depressive disorder with psychosis; those aged 36-45 years old must have had with onset of psychotic symptoms within the previous 5 years
* Achieved clinical stability, defined as outpatient status for at least one month prior to study participation

Exclusion Criteria:

* Unable or unwilling to provide informed consent
* The participant is unable to demonstrate adequate decisional capacity, in the judgment of the consenting study staff member, to make a choice about participating in the research study
* Participant is pregnant
* Participant is illiterate
* Cannot pass the CMRR Subject Safety Screen due to MRI contraindications
* Presence of a major neurological disorder (psychosis participants may have an autism spectrum diagnosis)
* Previous clinically significant head injury or prolonged unconsciousness, as determined by the PI/Co-Is
* Meets criteria for substance or alcohol dependence within 3 months of enrollment
* The presence of any major medical condition that, in the opinion of the PI/Co-Is, would impede participation in the study or would put the participant at additional risk by participating
* Presence of severe alcohol or substance abuse
* Has participated in significant formal cognitive training programs, as determined by the PI/Co-Is

Additional Exclusion Criteria for Early Psychosis Participants:

* Meets criteria for clinical risk of suicidal behavior, as defined by:
* Clinician judgement
* A suicide attempt within 6 months of enrollment
* Active suicidal ideation at screening or baseline, as indicated by the C-SSRS
* Previous intent to act on suicidal ideation with a specific plan and/or preparatory acts within 6 months of enrollment, as indicated by the C-SSRS

Additional Exclusion Criteria for Control Participants:

* Meets DSM-5 criteria for psychotic, bipolar, or autism spectrum disorder
* Has a family history (1st degree relative) of psychotic, bipolar, or autism spectrum disorder

Ages: 15 Years to 45 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult
Study Population: Participants are recruited from Minnesota. Most participants are located in the Twin Cities Metro area.
Sampling Method: Non-Probability Sample
Enrollment: 277 (Actual)
Dates: Start 2021-12-01 (Actual); Primary Completion 2025-08-29 (Actual); Study Completion 2025-08-29 (Actual)

PRIMARY OUTCOMES:
Change in Performance of Dot Pattern Expectancy (DPX) Task Variant | Baseline, 6 month follow up
  The DPX task variant consists of a series of pattern sequences. One pattern is designated the "A" cue, and another the "X" cue, which requires one response (AX, 60-70% of trials, e.g. respond with the left button), while other sequences require a different response (AY or BX, 12-15% of trials each, or BY, 6-10% of trials, e.g. respond with the right button). Given the strong expectation that X's evokes a valid response, BX trials place demands on the fidelity (stability, memory) of the "B" cue state representation to overcome this tendency. Performance is assessed based on accuracy and response time.
Change in Performance of Bandit Task Variant | Baseline, 6 month follow up
  This is a task variant that uses choice options (neutral images) that are rewarded probabilistically. The rewarded stimulus with the highest reward is changed over time. State learning associated with staying or switching stimuli too quickly (lose-switching) can be evaluated. Performance is based on accuracy, response time, and behavior of reward seeking.
Change in Test My Brain Neurocognitive Assessment performance: Global Cognition Z Score. | Baseline, 6 month follow up
  The investigators will examine global cognition scores from the Test My Brain neurocognitive battery. Z scores range from -5 to 5, with higher score indicating increased cognitive functioning.
Change in EEG Variables | Baseline, 6 month follow up
  Analysis will examine variables including phase synchrony, slope of the spectral power density (indexing E-I balance), and prefrontal/parietal theta as a measure of perceptual noise.
Change in MRI Variables | Baseline, 6 month follow up
  MRI assessments will include structural MRI, Diffusion-weighted MRI, Resting State fMRI.

SECONDARY OUTCOMES:
Change in symptoms and functioning as indicated by Minnesota Symptom Severity Scale | Baseline,6 month follow up
  This 29-item measure assesses symptoms in several domains such as anxiety, depression, sleep problems, somatic symptoms, and substance use. Scores range from 0 to 116, with a higher score indicating greater symptom severity.
Change in symptoms and functioning as indicated by the SANS/SAPS | Baseline, 6 month follow up
  The Scale for Assessment of Negative Symptoms (SANS, 25 items) and Scale for Assessment of Positive Symptoms (SAPS, 34 items) assess negative and positive symptoms of schizophrenia in a standardized interview. Scores on the SANS ranges from 0-125, and the SANS ranges from 0-170, with higher scores indicating increased symptom severity.
Change in symptoms and functioning as indicated by the BPRS | Baseline, 6 month follow up
  The Brief Psychiatric Rating Scale is a 24-item interview which assesses psychiatric symptoms. Scores on the BPRS rang from 24-168, with a higher score indicating increased symptom severity.
Change in symptoms and functioning as indicated by the SPQ-BR | Baseline, 6 month follow up
  Schizotypal Personality Questionnaire Brief Revised, a 32-item measure to assess a broad array of schizotypal symptoms and signs. The SPQ ranges from 32-160, with a higher score indicating greater schizotypy.
Change in symptoms and functioning as indicated by the SGI | Baseline, 6 month follow up
  The Sensory Gating Inventory Brief is a 10-item measure assesses an individual's subjective ability to modulate, filter, over-include, discriminate, attend to, and tolerate sensory stimuli. The SGI ranges from 10-60, with higher score indicating increased perceptual abnormalities.
Change in symptoms and functioning as indicated by the IDI | Baseline, 6 month follow up
  The Intersectional Discrimination Index is a 31-item measure assesses anticipated, day to day, and major discrimination experienced by the participant. Scores range from 0-136, with higher scores indicating greater discrimination experienced by the individual.
Change in symptoms and functioning as indicated by the WHODAS 2.0 Brief | Baseline, 6 month follow up
  The World Health Organization Disability Assessment Schedule is a 12-item self-administered scale measuring disability and functional impairment. The WHODAS ranges in score from 12-60, with a higher score indicating increased disability.
Change in symptoms and functioning as indicated by the GFS/GFR | Baseline, 6 month follow up
  The Global Functioning Social/Global Functioning Role scales provide a rating on a scale from 1-10 for social functioning and for role functioning, with higher scores indicating increased functioning.
Change in Test My Brain Neurocognitive Assessment performance: Digit Symbol Matching Z Score | Baseline, 6 month follow up
  This subdomain of the TMB battery assesses processing speed. Z scores range from -5 to 5, with higher score indicating increased functioning.
Change in Test My Brain Neurocognitive Assessment performance: Verbal Pair Associates Memory Z Score | Baseline, 6 month follow up
  This subdomain of the TMB battery assesses verbal learning. Z scores range from -5 to 5, with higher score indicating increased functioning.
Change in Test My Brain Neurocognitive Assessment performance: Matrix Reasoning Z Score | Baseline, 6 month follow up
  This subdomain of the TMB battery assesses reasoning skills and also provides an IQ estimate. Z scores range from -5 to 5, with higher score indicating increased functioning.
Change in Test My Brain Neurocognitive Assessment performance: Multiracial Emotion Identification Z Score | Baseline, 6 month follow up
  This subdomain of the TMB battery is a social cognition test that assesses the ability to recognize emotions (happiness, sadness, anger, and fear). Z scores range from -5 to 5, with higher score indicating increased functioning.

CONTACTS AND LOCATIONS:
Overall Officials: Sophia Vinogradov, MD, Principal Investigator — University of Minnesota; Angus MacDonald III, Ph.D., Principal Investigator — University of Minnesota
Locations (1):
- University of Minnesota, Minneapolis, Minnesota, United States

IPD SHARING:
Plan to Share IPD: Yes
This data is shared with the NIMH Data Archive, Collection ID C3504, and will include demographics, imaging data, and primary and secondary outcome data.
Supporting Information: Study Protocol, SAP
Time Frame: The data will become available 12 months after the completion of this study.
Access Criteria: Access will be provided to users who have an account with the NIMH Data Archive and who request permission through a Data Access Request.